CLINICAL TRIAL: NCT00594113
Title: Tailored Touch-Screens for Colorectal Cancer Prevention in Urban Core Clinics
Brief Title: "Touch 2 Screen" Multi-media Colorectal Cancer Screening Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allen A. Greiner, MD, MPH (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Allen A. Greiner, MD, MPH, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1RO1CA119098-01
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Multimedia Colorectal Cancer Screening
  Interventions: Other: Touch 2 Screen; Other: Touch screen intervention

INTERVENTIONS:
Other: Touch 2 Screen — Multi-media presentation and survey to increase screening for colorectal cancer. Content of this presentation is based on the concept of "implementation intentions," an advanced planning model taken from the Theory of Planned Behavior
Other: Touch screen intervention — Touch screen intervention

SUMMARY:
The primary purpose of this study is to determine the effectiveness of a multi-media presentation and survey to increase screening for colorectal cancer. Content of this presentation is based on the concept of "implementation intentions," an advanced planning model taken from the Theory of Planned Behavior. The multi-media presentation is delivered in a touch-screen computer format and contains messages about colorectal cancer that are tailored to each participant based on individual survey responses. It is hypothesized that tailored messages and defining implementation intentions may have a relationship with completion of colorectal cancer screening.

DETAILED DESCRIPTION:
The majority of the intervention will be delivered in primary care settings on low-cost touch-screen computers through multi-media audio-narrative and video messages. Studies have not tested the effectiveness of tailored communications specified to stated "implementation intentions" for improving CRC screening. A randomized design will test a comparison of generic information versus a multi-media tailored intervention that specifically addresses each participant's screening test preference, current CRC screening decisional state (Precaution Adoption Process Model), and specified to stated "implementation intentions" (the "when," "Where," and "how" details of screening.) Behavioral intervention materials in English and Spanish will be developed with the help of cultural experts, pilot tests, and interviews that will test salience and cultural appropriateness of audio, video, and graphic messages for low-income minorities and whites. The study will be conducted with 460 patients eligible for CRC screening and recruited while presenting for care in urban clinics. All participants will receive baseline touch-screen administered assessment and, depending on stated preference, be offered either immunochemical fecal occult blood test (iFOBT-InSureTM) or a colonoscopy. Participants will be randomized to either "C" (comparison group-computer delivered generic CRC information) or "TI2" (active intervention-computer delivered tailored messaging based on individual PAPM stage, behavioral constructs, and "implementation intentions"). A brief office exit survey will assess patient-provider discussions of CRC screening and satisfaction with computerized message materials. A 90-day post randomization follow-up telephone call assessment with all participants will reassess PAPM stage and perceived CRC screening barriers.

The primary outcome will be CRC screening completion at 90 days. Secondary outcomes will assess 90-day PAPM stage and perceived barriers among participants preferring various screening methods (iFOBT, Colonoscopy). This intervention will provide information on the utility of embedding a low-cost technologically advanced "implementation intentions" based behavioral intervention in primary care practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 50 years of age
* Must not have had a colonoscopy in the last 10 years
* Must not have completed Fecal Occult Blood Test in the past year
* Must not have a family history of colorectal cancer.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2007-08; Primary Completion 2010-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
CRC screening completion | 90 Days

SECONDARY OUTCOMES:
PAPM stage and perceived barriers among participants preferring various screening methods (iFOBT, Colonoscopy) | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Allen A. Greiner, MD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Background] Greiner KA, Geana MV, Epp A, Watson A, Filippi M, Daley CM, Engelman KK, James AS, Campbell M. A computerized intervention to promote colorectal cancer screening for underserved populations: theoretical background and algorithm development. Technol Health Care. 2012;20(1):25-35. doi: 10.3233/THC-2011-0653. PMID 22297711
- [Derived] Greiner KA, Daley CM, Epp A, James A, Yeh HW, Geana M, Born W, Engelman KK, Shellhorn J, Hester CM, LeMaster J, Buckles DC, Ellerbeck EF. Implementation intentions and colorectal screening: a randomized trial in safety-net clinics. Am J Prev Med. 2014 Dec;47(6):703-14. doi: 10.1016/j.amepre.2014.08.005. Epub 2014 Nov 18. PMID 25455115